CLINICAL TRIAL: NCT02267161
Title: Outcome of Infants With Prenatal Corpus Callosum Agenesis
Brief Title: Infants With Agenesis of the Corpus Callosum
Acronym: Dacci
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ID-RCB: 2014-A00625-42
Record Dates: First submitted 2014-07-17; First posted 2014-10-17 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Agenesis of the Corpus Callosum
Keywords: agenesis; corpus callosum; prenatal diagnosis
MeSH Terms: conditions — Agenesis of Corpus Callosum | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neuropsycological tests (Experimental): Psychometric scales for infants at 3 years of age
  Interventions: Other: Psychometric scales for infants at 3 years of age

INTERVENTIONS:
Other: Psychometric scales for infants at 3 years of age — WPPSI-III, VINELAND, CBCL, NEPSY

SUMMARY:
The purpose of this study is to assess the neurological development at three years of age of children born after prenatal diagnosis of "isolated" agenesis of the corpus callosum.

DETAILED DESCRIPTION:
Agenesis of the corpus callosum is the most frequent brain malformation. This anomaly may be diagnosed by ultrasound screening. In half of these prenatal cases, the anomaly seems to be isolated. In this setting, there are no prospective data concerning the development of these children, preventing any clear information to be delivered to parents. Prenatal diagnostic centers therefore face extremely variable rates of termination of pregnancies (TOP), which can reach up to 80%.

This is a multicentric prospective interventional study whose primary objective is to assess the neurological development at three years of age of children born after prenatal diagnosis of "isolated" agenesis of the corpus callosum.

Evaluation at three years will include Intellectual Quotient (IQ) quantification using the WPPSI-III, 3rd edition of Wechsler Preschool and Primary Scale of Intelligence and evaluation of intra-hemispheric coordination using the Vineland adaptative behaviour scale.

Secondary objectives will include:

* Circumstances leading to the prenatal diagnosis of agenesis of the corpus callosum
* Causes leading to termination of pregnancies
* Determination of criteria allowing to confirm that agenesis of the corpus callosum is isolated (family history, imagery, genetics)

These results could allow to determine the optimal prenatal management of such cases.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 28 weeks of gestation
* Complete agenesis of the corpus callosum
* Partial agenesis of the corpus callosum
* Abnormal corpus callosum (size, anatomy) As diagnosed by an expert ultrasound fetal brain examination.

Exclusion Criteria:

* age < 18 years old
* women who do not understand french
* women not covered by the French social security system
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-09-26 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
WPPSI-III (wechsler preschool and primary scale of intelligence) :evaluation of intellectual quotient ( questionnaire) | 3 years
  Neurodevelopment outcome

SECONDARY OUTCOMES:
Vineland adaptative behaviour scales (motricity capacity) : questionnaire | 3 years
  Neurodevelopment outcome
Nepsy : developmental neuropsychological assessment (capacity of coordination) | 3 years
  Neurodevelopment outcome
CBCL: Child Behavior Checklist (behaviour) : self administered questionnaire | 3 years
  Neurodevelopment outcome
Cerebral abnormalities | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Jouannic, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Armand Trousseau, Paris, France

REFERENCES:
- [Background] Sotiriadis A, Makrydimas G. Neurodevelopment after prenatal diagnosis of isolated agenesis of the corpus callosum: an integrative review. Am J Obstet Gynecol. 2012 Apr;206(4):337.e1-5. doi: 10.1016/j.ajog.2011.12.024. Epub 2011 Dec 27. PMID 22284958
- [Background] Moutard ML, Kieffer V, Feingold J, Lewin F, Baron JM, Adamsbaum C, Gelot A, Isapof A, Kieffer F, de Villemeur TB. Isolated corpus callosum agenesis: a ten-year follow-up after prenatal diagnosis (how are the children without corpus callosum at 10 years of age?). Prenat Diagn. 2012 Mar;32(3):277-83. doi: 10.1002/pd.3824. PMID 22430728
- [Background] Moutard ML, Kieffer V, Feingold J, Kieffer F, Lewin F, Adamsbaum C, Gelot A, Campistol I Plana J, van Bogaert P, Andre M, Ponsot G. Agenesis of corpus callosum: prenatal diagnosis and prognosis. Childs Nerv Syst. 2003 Aug;19(7-8):471-6. doi: 10.1007/s00381-003-0781-6. Epub 2003 Jul 4. PMID 12845459